CLINICAL TRIAL: NCT02757859
Title: The WASH Trial: A Randomized Trial of Abdominal Lavage Using Distilled Water or Saline at High Volumes for Resected Pancreatic Cancer
Brief Title: High Volume Washing of the Abdomen in Increasing Survival After Surgery in Patients With Pancreatic Cancer That Can Be Removed by Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16D.083; JT 6902 (Other: JeffTrial Number)
Record Dates: First submitted 2016-04-29; First posted 2016-05-02 (Estimated); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Acinar Cell Carcinoma; Ampulla of Vater Adenocarcinoma; Cholangiocarcinoma; Duodenal Adenocarcinoma; Pancreatic Adenocarcinoma; Pancreatic Ductal Adenocarcinoma; Pancreatic Intraductal Papillary Mucinous Neoplasm; Periampullary Adenocarcinoma
MeSH Terms: conditions — Carcinoma, Acinar Cell; Cholangiocarcinoma; Pancreatic Intraductal Neoplasms | interventions — Pancreatectomy; Therapeutic Irrigation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm I (EIPL-S) (Active Comparator): Patients undergo pancreaticoduodenectomy, distal pancreatectomy, or total pancreatectomy. Immediately after removal of tumor, patients receive EIPL-S lavage 10 times over 15 minutes.
  Interventions: Procedure: Pancreatectomy; Other: Lavage
- Arm II (EIPL-D) (Active Comparator): Patients undergo pancreaticoduodenectomy, distal pancreatectomy, or total pancreatectomy. Immediately after removal of tumor, patients receive EIPL-D lavage 10 times over 15 minutes.
  Interventions: Procedure: Pancreatectomy; Other: Lavage
- ARM III (NO LAVAGE) (Sham Comparator): Patients undergo pancreaticoduodenectomy, distal pancreatectomy, or total pancreatectomy with no extensive lavage after removal of tumor.
  Interventions: Procedure: Pancreatectomy

INTERVENTIONS:
Procedure: Pancreatectomy — Undergo pancreaticoduodenectomy, distal pancreatectomy, or total pancreatectomy
  Other Names: Excision of the Pancreas; Pancreas Excision
  Arms: Arm I (EIPL-S)
Other: Lavage — Receive EIPL-S
  Other Names: Irrigation; Wash
  Arms: Arm I (EIPL-S)
Procedure: Pancreatectomy — Undergo pancreaticoduodenectomy, distal pancreatectomy, or total pancreatectomy
  Other Names: Excision of the Pancreas; Pancreas Excision
  Arms: Arm II (EIPL-D)
Other: Lavage — Receive EIPL-D
  Other Names: Irrigation; Wash
  Arms: Arm II (EIPL-D)
Procedure: Pancreatectomy — Undergo pancreaticoduodenectomy, distal pancreatectomy, or total pancreatectomy
  Other Names: Excision of the Pancreas; Pancreas Excision
  Arms: ARM III (NO LAVAGE)

SUMMARY:
This randomized clinical trial studies how well high volume washing of the abdomen works in increasing survival after surgery in patients with pancreatic cancer that can be removed by surgery. High volume washings may remove free floating cancers present after surgery and help prolong survival in patients with pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Overall survival (OS) (18 to 27 months after resection).

SECONDARY OBJECTIVES:

I. Disease free survival (DFS). II. Complication rate. III. Site of first-recurrence (by site, and distant vs. local). IV. Clearance of malignant cells pre vs. post-lavage.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM I (EIPL-S): Patients undergo pancreaticoduodenectomy, distal pancreatectomy, or total pancreatectomy. Immediately after removal of tumor, patients receive extensive intraoperative peritoneal saline (EIPL-S) lavage 10 times over 15 minutes.

ARM II (EIPL-D): Patients undergo pancreaticoduodenectomy, distal pancreatectomy, or total pancreatectomy. Immediately after removal of tumor, patients receive extensive intraoperative peritoneal distilled water (EIPL-D) lavage 10 times over 15 minutes.

ARM III (NO LAVAGE): Patients undergo pancreaticoduodenectomy, distal pancreatectomy, or total pancreatectomy with no extensive lavage after removal of tumor.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a surgical indication for pancreatectomy (pancreaticoduodenectomy, distal pancreatectomy, total pancreatectomy) as determined by the treating physician/surgeon
* A diagnosis of pancreatic or other periampullary cancer is suspected preoperatively
* In the opinion of the surgeon, the subject has no medical contraindications to pancreatectomy
* Age ≥18 years of age.
* The subject is willing to consent to randomization of EAL-S vs. standard EAL-W vs. no extensive lavage. (SOC)

Exclusion Criteria:

* The subject does not have a surgical indication for pancreatectomy
* In the opinion of the surgeon, the subject has medical contraindications to pancreatectomy
* Age < 18 years of age
* The subject is not willing to consent to EAL-S vs. EAL-W vs. no extensive lavage (SOC)
* Known benign or indolent disease, including benign pancreatic cystic tumors or pancreatic endocrine tumors) without possible risk of malignancy
* Other malignancy within five years, unless the probability of recurrence of the prior malignancy is < 5% as determined by the principal investigator based on available information. Patient's curatively treated for squamous and basal cell carcinoma of the skin or patients with a history of malignant tumor in the past that have been disease free for at least five years are also eligible for this study.
* Evidence of metastatic disease preoperatively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 845 (Estimated)
Dates: Start 2016-04-27 (Actual); Primary Completion 2026-04-27 (Estimated); Study Completion 2026-04-27 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Up to 27 months after resection
  Will use a one-sided log-rank test to separately compare lavage (EIPL-S or EIPL=D) to no lavage with respect to OS. Assuming the study is not stopped at the interim analyses, the final comparison will be made with an alpha level of 0.02493. Distribution of OS will be estimated using the Kaplan-Meier method. Secondary analyses will use Cox regression to adjust the lavage/no lavage comparison for other baseline patient and/or characteristics known to be associated with OS.

SECONDARY OUTCOMES:
Incidence of overall complications and specific complications graded in severity using Common Terminology Criteria for Adverse Events (v4.0) | Up to 5 years after resection
  Will use chi-square or Fisher's exact test for dichotomous outcomes and Poisson regression for count outcomes.
Disease Free survival | Up to 5 years after resection
  Will use log-rank tests for time-to-event outcomes.
Recurrence free survival rate | At 1 year after resection
Site of first recurrence | Up to 5 years after resection

OTHER OUTCOMES:
Presence of cells in cytologic washing | Up to 5 years
  Will be modeled with repeated measures logistic regression using generalized estimating equations methods. Within this model, group differences in change from post-resection to post-lavage will be compared. McNemar's test for paired dichotomous data will be used to compare presence of cells at pre-dissection to post-resection.

CONTACTS AND LOCATIONS:
Overall Officials: Harish Lavu, MD, Principal Investigator — Thomas Jefferson University
Locations (2):
- United States (2):
  - Case Western Reserve University, Cleveland, Ohio
  - Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/